CLINICAL TRIAL: NCT01091285
Title: Induction of Labor With Single and Double Balloon Catheters, a Randomized Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Birte Haugland, Dr, Womens hospital, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1728a (REK)
Record Dates: First submitted 2010-03-20; First posted 2010-03-24 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2010-04

CONDITIONS: Induction of Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Single Balloon Catheter (Active Comparator): Cervix Ripening is achieved by a single balloon catheter. Further induction by cytotec or/amniotomy and pitocin
  Interventions: Device: Foley Catheter
- Double balloon catheter (Active Comparator): Cervix Ripening is achieved by a double balloon catheter. Further induction by cytotec or/amniotomy and pitocin
  Interventions: Device: Double Balloon Catheter

INTERVENTIONS:
Device: Foley Catheter — Foley Catheter 16-19 H
  Arms: Single Balloon Catheter
Device: Double Balloon Catheter — Double Balloon Catheter for 16-19H
  Other Names: Cervical Ripening Balloon, Cook Medical
  Arms: Double balloon catheter

SUMMARY:
A randomized controlled double blinded study to investigate whether a specially designed double balloon catheter is more efficient than a foley catheter for cervical ripening and induction of birth.

160 women with singleton term pregnancies with un ripe cervix and no contraindications for catheters will be included and randomized to either double og single balloon catheters for cervical ripening. Efficacy wil be assessed at removal of the catheter, measured by the amount of women where the cervix has become ripe enough for amniotomy.

Our hypothesis is that double balloon catheters will give a greater amount of women where amniotomy upon catheter removal is possible. Secondary outcomes as time from induction till birth, vaginal deliveries and complications during or after birth for the mother or child will also become recorded.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy above week 37
* Indication to induce birth
* Unripe cervix
* Term date set by US before week 21

Exclusion Criteria:

* Ripe cervix
* Prematurity (<37w)
* IUFD
* Letal malformations
* Low lying placenta
* Multiple pregnancies
* Breakage of amniotic fluid
* The woman does not understand norwegian

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Cervix dilatation >= 3cm | At cather removal
  Cervix dilatation is assessed by vaginally examination at Catheter removal.

CONTACTS AND LOCATIONS:
Locations (1):
- Womens Hospital, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264